CLINICAL TRIAL: NCT03148782
Title: Brain Plasticity Underlying Acquisition of New Organizational Skills in Children
Brief Title: Brain Plasticity Underlying Acquisition of New Organizational Skills in Children-R61 Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R61/17-00263; R61MH113663 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder; Neurodevelopmental Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OST Intervention (Experimental): 12 weekly in-person sessions, each lasting approximately 1 hour, targeting 3 core organizational skills domains-Tracking Assignments, Managing Materials and Time Management
  Interventions: Behavioral: OST Intervention for participants with Organizational skill difficulties

INTERVENTIONS:
Behavioral: OST Intervention for participants with Organizational skill difficulties — Will undergo two magnetic resonance imaging (MRI) sessions: one within 2 weeks prior to OST treatment and one within 2 weeks of completion of the OST treatment.

SUMMARY:
Organizational, time management and planning (OTMP) skills deficits are seriously impairing features of developmental disorders, such as Attention Deficit Hyperactive Disorder (ADHD) and autism, which compromise school performance and family relations. The manualized Organizational Skills Training program (OST) was designed to target children's specific OTMP deficits. However, the brain mechanisms of treatment-induced changes remain unknown. The current study combines a training intervention with non-invasive MRI imaging in a pre-/post-design to address this question.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry: age ≥ 8.0 and ≤ 11.9 years corresponding to grades 3-5
* Written assent by child and consent by parent or legal guardian
* IQ: Estimated full scale IQ ≥ 85 and language comprehension scores ≥ 80 is required as in past studies to assure that children are able to comply with specific skills training and to minimize neurobiological heterogeneity
* Organizational skills deficits defined as elevated (≥ 1SD) pre-treatment COSS Parent Total T-score and at least one COSS Parent Interference item rated as either a 3 or 4 (indicating an above-average level of impairment)
* Handedness: given the greater prevalence of non-right-handedness in neurodevelopmental disorders, we will track handedness but not exclude left-handed individuals
* Medication: To minimize variability due to medication effects, we will preferentially recruit currently unmedicated individuals (no psychoactive medications in the previous 3 months). For stimulants, we will require that dosage be stable for >1 month before study entry and parents will be asked to consult their physician regarding discontinuation for 48 hours before evaluation, mock scanning and scanning sessions.
* Must provide adequate MRI data at baseline

Exclusion Criteria:

* Enrolled in a self-contained special education classroom or served by a 1:1 paraprofessional in their classroom
* A learning disability on Individualized Education Plan
* Absence of signed consent by parent or legal guardian
* Children who dissent regardless of parental permission
* Full scale IQ < 85
* Participants for whom stimulant discontinuation for 48 hours prior to evaluation, mock scan and scanning sessions is deemed medically impermissible
* Children with a recent (past 6 months) or current history of neuroleptic treatment or current treatment with psychotropic medications other than stimulants
* Per history (and medical records if needed) medical illness requiring chronic current treatment
* History of intrathecal chemotherapy or focal cranial irradiation
* Premature birth (< 32 weeks estimated gestational age or birth weight < 1500g)
* History of leukomalacia or static encephalopathy, intracerebral hemorrhage beyond grade 2, other specific or focal neurological or metabolic disorder including epilepsy (except for resolved febrile seizures)
* History of traumatic brain injury
* Contraindication for MRI scanning (metal implants, pacemakers, metal foreign bodies or pregnancy)

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in parent Children's Organizational Skills Scales (COSS-P) total T-scores following OST intervention. | Day 1
  Parents (COSS-P) and teachers (COSS-T) will serve as informants (only the child is a study subject) who will provide baseline and outcome ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco X Castellanos, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be provided to the National Database for Clinical Trials Related to Mental Illness (NDCT) for sharing to other researchers.